CLINICAL TRIAL: NCT02727959
Title: Inflammatory Bowel Disease in South Eastern Norway (IBSEN III). Clinical Epidemiology, Diagnostic and Prognostic Factors in Inflammatory Bowel Disease.
Brief Title: Inflammatory Bowel Disease in South Eastern Norway
Acronym: IBSENIII
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other); Oslo Metropolitan University (Other); Takeda (Industry); Ferring Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Marte Lie Høivik, MD Postdoc PhD, Oslo University Hospital
Other Study IDs: 581912
Record Dates: First submitted 2016-02-15; First posted 2016-04-05 (Estimated); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Colitis, Ulcerative; Crohn Disease; Inflammatory Bowel Disease
Keywords: UC; CD; IBD
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients newly diagnosed with IBD
- Symptomatic non IBD-controls: Patients referred with symptoms suspicious of IBD, but who, after examination, are found not to have the diagnosis.

SUMMARY:
The IBSEN III study will investigate the incidence of inflammatory bowel disease in South Eastern Norway and describe the clinical course of the disease. The investigators will map newly diagnosed and treatment naive IBD patients at various levels (epidemiological, clinical, psychosocial and nutritional as well as immunological, genetic, epigenetic and microbial) as a basis to improve targeted and individualized treatment and care. The investigators will include incident IBD patients at all local- and university hospitals in the South Eastern Health Region in 2016-2018 and follow-up prospectively for five years. The investigators will use standardized and validated registration methods allowing comparability with previous national and international IBD cohorts, link data to national health registries and collect blood, feces and biopsies for bio banking.

ELIGIBILITY:
Inclusion Criteria:

Ulcerative colitis:

Diagnostic criteria (at least three out of four criteria present):

1. A history of diarrhea and/or pus in stools for more than 4weeks or repeated episodes.
2. Macroscopic appearance at endoscopy of continuous mucosal inflammation affecting the rectum in continuity with some or the entire colon.
3. Microscopic features on biopsy compatible with UC,
4. No suspicion of CD on small bowel X-ray, ileocolonoscopy or biopsy.

Crohn's disease:

Diagnostic criteria (at least two of four criteria present):

1. History of abdominal pain, weight loss and/or diarrhea for more than three months.
2. Characteristic endoscopic findings of ulceration (aphthous lesions, snail track ulceration) or cobble stoning or radiological features of stricture or cobble stoning.
3. Histopathology consistent with Crohn's disease (epitheloid granuloma of Langerhans type or transmural discontinuous focal or patchy inflammation).
4. Fistula and/or abscess in relation to affected bowel segments.

Inflammatory bowel disease, type unclassified (IBDU) :

Patients with evidence on clinical and endoscopic grounds for chronic inflammatory bowel disease affecting the colon, without small bowel involvement, and no definitive histological or other evidence to favor either CD or UC.

Pediatric patients:

Will be diagnosed according to the Porto-criteria and defined as:

Pediatric onset IBD ≤ 16 years Early Onset IBD (EOIBD) < 10 years Very Early Onset IBD (VEOIBD) < 6 years Infantile (and toddler) IBD < 2 years Neonatal IBD < 28 days

Exclusion criteria:

* Other causes of acute or chronic bowel inflammation must be excluded, i.e. infectious colitis, radiation colitis, diversion colitis, solitary rectal ulcer syndrome, graft versus host disease, diverticular colitis, medication associated colitis, ischemic colitis, microscopic colitis, enema associated colitis.
* Refusal or not able to give informed consent

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult and pediatric patients untreated and newly diagnosed with inflammatory bowel disease i.e ulcerative colitis or Crohns disease as well as non-IBD Controls.
Sampling Method: Non-Probability Sample
Enrollment: 2286 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Evidence for ulcerative colitis, Crohn's disease or indeterminate colitis based on specific clinical, endoscopic, histological and radiological criteria | At baseline
  Diagnosis according to the Lennard Jones Criteria for the diagnosis of inflammatory bowel disease

SECONDARY OUTCOMES:
Change in IBD diagnosis between baseline and one year follow-up | 1 year (+/-3 months)
  Change in diagnosis based on specified clinical, endoscopic, histological and radiological criteria
Change in IBD diagnosis between one year and five year follow-up | 5 year (+/-3 months)
  Change in diagnosis based on specified clinical, endoscopic, histological and radiological criteria
Change in disease classification (montreal Classification) between baseline and one year follow-up. | 1 year (+/-3 months)
  Change in disease extension and severity as defined in the Montreal classification system for IBD
Change in disease classification (montreal Classification) between one and five year follow-up | 5 year (+/-3 months)
  Change in disease extension and severity as defined in the Montreal classification system for IBD
IBD related bowel surgery | 1 year (+/-3 months)
  Bowel surgery for any IBD related condition
IBD related bowel surgery | 5 year (+/-3 months)
  Bowel surgery for any IBD related condition

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Andersen S, Bernklev T, Stordal K, Hagen MC, Kristensen VA, Opheim R, Olbjorn C, Rove J, Lovlund EE, Holm HK, Aballi B, Hoivik ML, Perminow G. Specific phenotypes may drive an increased incidence of pediatric inflammatory bowel disease in South-Eastern Norway. J Pediatr Gastroenterol Nutr. 2025 Nov;81(5):1227-1236. doi: 10.1002/jpn3.70148. Epub 2025 Sep 1. PMID 40888250
- See also: IBSEN III webpage — https://www.med.uio.no/klinmed/english/research/projects/ibsen-inflammatory-bowel-disease/